CLINICAL TRIAL: NCT06151379
Title: The Relation Between the Initial Value of the Skeletal Mass Index and Pathological Response
Brief Title: Muscle Parameters and Pathological Response in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Acıbadem Atunizade Hospital (Other)
Responsible Party: Principal Investigator, Ebru Yilmaz, Principal Investigator, Acıbadem Atunizade Hospital
Other Study IDs: AcıbademAH
Record Dates: First submitted 2023-11-04; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Neoadjuvant Chemotherapy
Keywords: operable breast cancer; skeletal mass index; neoadjuvant chemotherapy; pathologic response; L3 vertebra
MeSH Terms: interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pathologic complete response (pCR): Patient with complete pathological response
  Interventions: Other: Neoadjuvant therapy
- Pathologic incomplete response (non-pCR): Patient with partial pathological response
  Interventions: Other: Neoadjuvant therapy

INTERVENTIONS:
Other: Neoadjuvant therapy — To measure muscle mass and predict pCR to NAC and its effect on clinical outcomes.

SUMMARY:
The investigators aimed to accurately measure muscle mass and predict pCR to NAC and its effect on clinical outcomes.

DETAILED DESCRIPTION:
In patients with operable breast cancer (BC) receiving neoadjuvant chemotherapy (NAC), the pathological response rate was found to be related to body composition. The success of complete pathologic response (pCR) is a known prognostic factor in BC patients treated with NAC. The investigators aimed to accurately measure muscle mass and predict pCR to NAC and its effect on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Early and locally advanced operated breast cancer patients receiving neoadjuvant chemotherapy.

Exclusion Criteria:

* Patients who did not receive neoadjuvant chemotherapy, had metastatic breast cancer and whose radiological images were not available.

Ages: 29 Years to 72 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Early and locally advanced operated breast cancer patients receiving neoadjuvant chemotherapy.
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Sarcopenic index | Through study completion, an average of 1 year.
  skeletal muscle area (cm2)/height (m2) et L3 level

SECONDARY OUTCOMES:
Body mass index | Through study completion, an average of 1 year.
  weight (kg)/height (m2)

OTHER OUTCOMES:
Residual cancer burden | Through study completion, an average of 1 year.
  Residual cancer burden (RCB) is estimated from routine pathologic sections of the primary breast tumor site and the regional lymph nodes after the completion of neoadjuvant therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Aysun Isiklar, M.D., Principal Investigator — Acıbadem Atunizade Hospital
Locations (1):
- AcıbademAH, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No